CLINICAL TRIAL: NCT05843565
Title: Standard Versus Hyperangulated Video Laryngoscopy Blades for Intubation in Neonates and Small Infants: Evaluation of the Glottic View
Brief Title: Standard Versus Hyperangulated Video Laryngoscopy Blades for Intubation in Neonates and Small Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Marie Awad, Principal investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2022-0348
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Intubation; Difficult or Failed
Keywords: Intubation; Laryngoscopy; Pediatrics; Neonates

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence of NSB first (Experimental): In patients allocated to the sequence of NSB first, the POGO and C&L classification will be recorded using video laryngoscopy with the hyperangulated blade 2 followed by an assessment using the Miller blade 0 or 1. Intubation will then be attempted during the second assessment. Endotracheal tube size will be selected according to body weight and a guiding stylet will be used. If the first attempt at intubation fails, the subsequent attempts will be left at the discretion of the attending anesthesiologist.
  Interventions: Device: Non-standard blade (NSB); Device: Standard blade (SB)
- Sequence of SB first (Placebo Comparator): In patients allocated to the Miller group, the POGO and C&L classification will be recorded using video laryngoscopy with a Miller blade 0 or 1 followed by an assessment using the Cobalt blade 2. Intubation will then be attempted during the second assessment. Endotracheal tube size will be selected according to body weight and a guiding stylet will be used. If the first attempt at intubation fails, the subsequent attempts will be left at the discretion of the attending anesthesiologist.
  Interventions: Device: Non-standard blade (NSB); Device: Standard blade (SB)

INTERVENTIONS:
Device: Non-standard blade (NSB) — GlideScope® VL (Verathon Inc, WA, USA) hyperangulated blade 2
Device: Standard blade (SB) — standard Miller blade 0 or 1

SUMMARY:
The goal of this prospective randomized cross over clinical trial is to compare the difference in the percentage of glottic opening (POGO) between two different video laryngoscopy blades, the hyperangulated Cobalt blade and the straight Miller blade in neonates or small infants with body weight ≤ 5 kg and age ≤ 3 months.

The main questions it aims to answer are:

* Is there a significant difference in the POGO using the standard Miller video laryngoscope blade versus the non-standard hyperangulated Cobalt video laryngoscope blade in neonates and small infants?
* Are there significant differences in the first attempt success rate at intubation, the number of attempts, the time to successful intubation, the type of blade used for successful intubation, and the occurrence of adverse events during intubation, such as episodes of bradycardia or desaturation?

  40 (20 in each group) neonates or small infants with body weight ≤ 5 kg or age ≤ 3 months will be enrolled in one of the two groups over 2 years of work.

Researchers will compare the POGO and Cormack and Lehane (C&L) classification using the hyperangulated Cobalt blade versus the straight Miller blade to identify the technique that provides optimal glottic views and intubating conditions in this patient population, and thus improved patient's safety.

DETAILED DESCRIPTION:
A higher incidence of difficult airway has been reported in neonates and infants than in adults. Optimizing glottic view during tracheal intubation is very challenging in neonates and small infants and it is not clear whether the design of the intubating blade using video laryngoscopy has a major influence of the glottic view and subsequently on the success of intubation.

The primary objective of this study is to compare the difference in the percentage of glottic opening (POGO) between two different video laryngoscopy blades, the hyperangulated Cobalt blade and the straight Miller blade. The secondary objectives are the first attempt success rate at intubation, the number of attempts, the time to successful intubation, and the occurrence of adverse events during intubation, such as desaturation or bradycardia.

In this prospective randomized cross over clinical trial, 40 (20 in each group) neonates or small infants with body weight ≤ 5 kg or age ≤ 3 months will be enrolled in one of two groups over 1 year of work. In patients allocated to the Cobalt group, the POGO and Cormack and Lehane (C&L) classification will be recorded using video laryngoscopy with a Cobalt blade followed by an assessment using the Miller blade. In patients allocated to the Miller group, the POGO and C&L classification will be recorded using video laryngoscopy with a Miller blade followed by an assessment using the Cobalt blade. In both groups, intubation will be attempted during the second assessment. If the first attempt at intubation fails, the subsequent attempts will be left at the discretion of the attending anesthesiologist.

Data comparing straight and hyperangulated video laryngoscopy blades in neonates and small infants are limited. Both techniques are standard of care at our institution. This study will identify the technique that provides optimal glottic views and intubating conditions in this patient population, and thus improved patient's safety.

ELIGIBILITY:
Inclusion Criteria:

* Neonates or small infants with body weight ≤ 5 kg or age ≤ 3 months, scheduled for elective surgery under general anesthesia.
* ASA (American Society of Anesthesiologists) class I-III patients.

Exclusion Criteria:

* Patients with a history of difficult airway or with craniofacial and airway anomalies.
* ASA (American Society of Anesthesiologists) class IV patients.
* Recent respiratory tract infection within the last 2 weeks.

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
POGO % | Intraoperatively
  Percentage of Glottic Opening
C&L classification | Intraoperatively
  Cormack and Lehane classification for glottic view.

SECONDARY OUTCOMES:
Intubation attempts | Intraoperatively
  Number of intubation attempts.
Time to successful tracheal intubation | Intraoperatively
  Anesthesia timeline (seconds) from first intubation attempt to first EtCO2 detection
Adverse events during intubation | Intraoperatively
  Occurrence of events such as: Desaturation (SpO2 < 95%) and bradycardia.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Aouad-Maroun, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No